CLINICAL TRIAL: NCT01034618
Title: The Additional Effects of Protein Hydrolysate Supplementation on Glucose Homeostasis in Type 2 Diabetes
Brief Title: Protein Hydrolyzation and Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Ralph J.F. Manders, PhD, Maastricht University Medical Center
Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 06-3-081
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes
Keywords: Diabetes; protein; protein hydrolysate
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Protein hydrolyzation
- Intact protein (Experimental)
  Interventions: Dietary Supplement: Protein hydrolyzation
- Protein hydrolysate (Experimental)
  Interventions: Dietary Supplement: Protein hydrolyzation

INTERVENTIONS:
Dietary Supplement: Protein hydrolyzation

SUMMARY:
The insulinotropic effects of protein hydrolysate/amino acid ingestion have been shown to regulate blood glucose homeostasis in both type 2 diabetes patients and normoglycemic controls. The objective of the study is to investigate the optimal dose of such an insulinotropic mixture.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 40 and 70 years
* Oral blood glucose lowering medication
* BMI < 35 kg/m2

Exclusion Criteria:

* Exogenous insulin use
* Cardiac disease (any cardiac event in the last 5 years)
* Diabetic complications (microvascular complications, microalbuminuria: albumin:creatinine ratio >2,5)

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Glucose and insulin homeostasis.

SECONDARY OUTCOMES:
Plasma amino acid profiles

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands